







## **SYNOPSIS APPAHOCA study**

Feasibility of adapted physical activity based on a walking platform for elderly patients hospitalized for cancer

**ID-RCB: 2018-A00031-54** Version n°2.1 07/10/2018

| SPONSOR | Centre François Baclesse 3 avenue du Général Harris 14076 CAEN cedex 5 | |
|---|---|---|
| COORDINATING<br>INVESTIGATORS | Dr Bérengère BEAUPLET CHU - Avenue Côte de Nacre 14033 CAEN Cedex Dr Heidi SOLEM LAVIEC Centre François Baclesse Boulevard du Général Harris 14000 CAEN | |
| REGULATORY<br>APPROVALS | CPP IDF 5 | Date: 06/03/2018 |

| TITLE | Feasibility of adapted physical activity based on a walking platform for elderly patients hospitalized for cancer |
|---|---|
| ACRONYM | АРРАНОСА |
| Coordinator | Dr Bérengère BEAUPLET |
| Indication | Elderly patients hospitalized for cancer |
| Test<br>methodology | Multicenter, prospective, non-randomized, open-label pilot feasibility study |
| | Main objective |
| Objectives | Assess the feasibility of adapted physical activity (APA) based on a walking platform in patients aged 70 and over hospitalized for cancer. Secondary objectives |
| | <ul> <li>Describe adherence to adapted physical activity, in quantitative and qualitative terms</li> <li>Investigate factors associated with adherence: oncological factors, social factors, previous mobility, cognitive level, comorbidities</li> <li>Assess patient satisfaction with using an adapted walking platform</li> </ul> |
| | Main criteria |
| | <ul> <li>Percentage of patients included who complete at least two sessions of 6 minutes or more of adapted physical activity on the walking platform.</li> <li>Adapted physical activity on a walking platform will be considered feasible if ≥70% of patients complete ≥2 sessions of 6 minutes or more during their hospitalization for cancer lasting ≥48 hours.</li> <li>Secondary criteria</li> </ul> |
| | Patient adherence to adapted physical activity will be assessed: • Quantitatively (intensity of participation): number and duration of sessions, number and regularity of steps, maximum and average walking speed, distance covered • Qualitatively: o Reason for not completing the first and/or second session, o Type of activity: use of balance games, chosen visual walking route |
| Judgment<br>criteria | Factors that may be associated with adherence: Gender, age, socio-professional category before retirement Location of cancer, reasons for hospitalization (medical or surgical) Pain Activity before hospitalization: Performance Status, previous QAPPA activity level, history of falls in the past year Cognitive status prior to the first session: memory test (temporal-spatial orientation/10, learning and recalling 3 words) Activity prior to the first session: Ability to walk 4 meters (alone/with technical and/or human assistance) and time required; Ability to transfer (alone/with technical and/or human assistance); Physical therapy already underway Context, presence of severe comorbidity(ies) affecting mobility, presence of isolation due to multi-resistant bacteria, presence of medical equipment (IV, drain, urinary catheter, enteral feeding tube, ostomy bag, oxygen therapy glasses) Patient satisfaction with the use of the adapted walking platform will be assessed at each session on a scale of 0 to 10 on the following items: |

| | 1 11 60 1 10 |
|---|---|
| | <ul><li> Use of the treadmill</li><li> Satisfaction with the digital tablet on the walking platform</li></ul> |
| | <ul> <li>Instructional support from the APA educator (starting from the second<br/>session)</li> </ul> |
| Inclusion<br>criteria | - Patients with cancer |
| | - Patients over the age of 70 hospitalized for 48 hours or more |
| | - Patients identified as eligible for a medical prescription for APA |
| | - Proficiency in French |
| | - Patients affiliated with a social security system |
| | - Patients who have given their written consent |
| Exclusion<br>criteria | - Patients who are completely unable to communicate |
| | - Patients receiving palliative care in the terminal phase |
| | - Patients who are less than 1.35 m or more than 2 m tall and/or weigh more than 130 kg |
| | - Patients who are unable to participate in APA sessions |
| | - Patients who are unable to wear a support harness |
| | - Patients deprived of their liberty or under guardianship |
| | <ul> <li>Patients unable to comply with the requirements of the protocol for<br/>geographical, social, or psychopathological reasons</li> </ul> |
| Description of the | After checking the patient's ability to participate in walking sessions and obtaining a medical prescription, the physical activity instructor will ask patients questions about their usual activities prior to hospitalization. |
| | During the patient's hospitalization, physical activity on the adapted ema® walking platform will be offered every working day, in the form of a session lasting a minimum of 6 minutes and a maximum of 30 minutes. |
| protocol/exp<br>erimental | The walking sessions will be carried out on an adapted walking platform, comprising a treadmill and a connected tablet. The tablet allows patients to view a landscape or |
| design | play balance or memory games while walking. The activity offered will be tailored to the patient's profile. |
| | Patients will be brought to the platform in a wheelchair and returned to their room by the same means of transport. |
| | At the end of each session, patients will complete a satisfaction questionnaire. |
| Number of subjects | To estimate a proportion of 70% of patients with a 95% confidence interval of [45-95], it is necessary to include 50 evaluable patients. To anticipate potential non-evaluable patients, we plan to include 60 patients. |
| Participating centers | 2 |
| Study<br>duration | 6 months |